CLINICAL TRIAL: NCT05228405
Title: Awareness Levels of Caregivers of Disabled Children About Children's Illness, Physiotherapy and Sports Activities
Brief Title: Awareness Levels of Caregivers of Disabled Children
Acronym: caregivers
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Assistant Proffessor, Kahramanmaras Sutcu Imam University
Other Study IDs: KSU5
Record Dates: First submitted 2022-01-23; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Cerebral Palsy; Caregiver Burden; Disabilities Multiple; Muscular Dystrophy; Down Syndrome; Spina Bifida
Keywords: awareness, caregiver, disabled, physiotherapy, sports
MeSH Terms: conditions — Cerebral Palsy; Caregiver Burden; Muscular Dystrophies; Down Syndrome; Spinal Dysraphism | interventions — Physical Therapy Modalities; Weights and Measures

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/caregivers of disabled children: 1/Caregivers of disabled children will be assessed by the questionnaire of the Disease, Physiotherapy and Sports Awareness
  Interventions: Other: All of the disabled children's caregivers will answer the Questionnaire of Disease, Physiotherapy and Sports Awareness

INTERVENTIONS:
Other: All of the disabled children's caregivers will answer the Questionnaire of Disease, Physiotherapy and Sports Awareness — All of the different type of disabled children's caregivers (cerebral palsy, muscular dystrophy, spina bifida and down syndrome) will answer the Questionnaire of Disease, Physiotherapy and Sports Awareness
  Other Names: scale

SUMMARY:
Disability-or apology; It is the inability or incompleteness of individuals to fulfill their roles in life, such as age, gender, culture, social and psychological factors, due to their inadequacies. Disability is not only a mental or physical health problem, but also a social problem. Having a disabled child and the type of disability present various difficulties to parents in the course of life. The difficulties in the care and education of these children are based on psychological, physical, social, economic and cultural realities.Families with diseases such as Cerebral Palsy (SP), Spina Bifida (SB), Muscular Dystrophy (MD), Down Syndrome (DS) are among them. Having a disabled child in the community can affect families in different ways. Every step of the education of disabled children (purpose, principle, education plan, game, school and family duties, etc.) is important for the disabled individual, family, teacher and society.

DETAILED DESCRIPTION:
Parents spare more time for the care and health of their disabled children, limited time spent with other family members, families do not have much information about their children's disabilities after the diagnosis of disability, limited life in children's vision, hearing, speech, mental and physical activities, functional losses this increases the difficulties. Self-care problems such as sleeping, eating, drooling, inactivity and dressing skills in children with CP, difficulties experienced by children with mental disabilities in making friends and acting independently, problems in going to school, financial losses during the creation of an environment and environment suitable for their disability, frequently They face many difficulties such as adaptation problems and behavioral problems, and the perspective that society has formed against them due to their differences in body characteristics. As the life span of people with disabilities increases, the financial, moral, physical and social difficulties of their families increase, and over time, psychological and behavioral barriers occur in family members. These barriers are increasing in developing countries. Social support is one of the most important factors that facilitate successful adaptation to the presence of a child with a disability and reduce the level of stress they feel in their lives. Social support refers to the help an individual receives from other people. It can be defined as information that enables a person to have the belief that they are loved, valued, accepted and part of an interpersonal support network. Individuals can receive social support from their spouse, family and friends, as well as from leisure activities, recreational activities, community programs, and professionals and institutions. Social support or the perception of social support plays an important role in maintaining the mental health of families. Studies on social support show that as social support of individuals with disabled children increases, their psychological symptoms, hopelessness levels, depressive symptoms and stress levels decrease; revealed that their adjustment and well-being increased. Küçükahmet stated that the institutions in that society have an impact on the upbringing and development of children in every society and that one of these institutions is the family.Today, it is known that family-centered approaches are the most successful in terms of rehabilitation of individuals with disabilities. Because it is known that the family is of great importance in terms of ensuring the active participation of the child in life. Therefore, while interdisciplinary treatments continue for the treatment of individuals, the success of rehabilitation depends on interacting with the family, identifying and supporting their needs and problems. For this reason, with this study, it is planned to investigate whether the parents know enough about the physiotherapy program applied to their children, what level of knowledge they have about their children's disease, and whether their disabled children participate in sports activities. The aim of this study is to measure the level of awareness of parents with disabled children about disease, physiotherapy and sports.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of children with GMFCS Level (Gross Motor Function Classification System) 1-4, aged 4-20, with Cerebral Palsy (SP), Spina Bifida (SB), Down syndrome (DS) and Muscular Dystrophy (MD) diseases
* Voluntary participating parents who live in Gaziantep and have a child with one of the selected disease groups

Exclusion Criteria:

* Parent has any diagnosed mental illness

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Caregivers of children with GMFCS Level (Gross Motor Function Classification System) 1-4, aged 4-20, with Cerebral Palsy (SP), Spina Bifida (SB), Down syndrome (DS) and Muscular Dystrophy (MD) diseases
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Questionnaire of Disease, Physiotherapy and Sports Awareness (QODPSA) (for cerebral palsy) | first day of assessment
  All of the caregivers of the different disabled children will be assessed by the Questionnaire of Disease, Physiotherapy and Sports Awareness(QODPSA). There are questions for the parents of the children of the cerebral palsy. This questionnaire has only one correct answer. Survey questions are multiple choice. The content of the survey questions; consists of diseases, physiotherapy and sports. Higher scores on this scale indicate better awareness levels.
Questionnaire of Disease, Physiotherapy and Sports Awareness (QODPSA) (for muscular dystrophy) | first day of assessment
  All of the caregivers of the different disabled children will be assessed by the Questionnaire of Disease, Physiotherapy and Sports Awareness(QODPSA). There are questions for the parents of the children of the muscular dystrophy in this questionnaire. This questionnaire has only one correct answer. Every survey questions are multiple choice. The questionnaire consists of diseases, physiotherapy and sports. Higher scores on this scale indicate better awareness levels.
Questionnaire of Disease, Physiotherapy and Sports Awareness (QODPSA) (for spina bifida) | first day of assessment
  All of the caregivers of the different disabled children will be assessed by the Questionnaire of Disease, Physiotherapy and Sports Awareness(QODPSA). There are questions for the parents of the children of the spina bifida in this questionnaire. This questionnaire has only one correct answer. Every survey questions are multiple choice. The questionnaire consists of diseases, physiotherapy and sports. Higher scores on this scale indicate better awareness levels.
Questionnaire of Disease, Physiotherapy and Sports Awareness (QODPSA) (for down syndrome) | first day of assessment
  All of the caregivers of the different disabled children will be assessed by the Questionnaire of Disease, Physiotherapy and Sports Awareness(QODPSA). There are questions for the parents of the children of the down syndrome in this questionnaire. This questionnaire has only one correct answer. Every survey questions are multiple choice. The questionnaire consists of diseases, physiotherapy and sports. Higher scores on this scale indicate better awareness levels.

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No